CLINICAL TRIAL: NCT04907825
Title: A Trial of Pharmacist Management of Oral Anticoagulation THerapy Versus Enhanced Usual CARe in the communitY for AF (APOTHECARY AF Study)
Brief Title: A Trial of Pharmacist Management of Oral Anticoagulation THerapy Versus Enhanced Usual CARe in the communitY for AF
Acronym: APOTHECARYAF
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Roopinder Sandhu, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00000850
Record Dates: First submitted 2021-05-13; First posted 2021-06-01 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: Atrial Fibrillation; Stroke; Oral Anticoagulants; Pharmacist Case Management
MeSH Terms: conditions — Atrial Fibrillation; Stroke | interventions — Anticoagulants; Warfarin

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, cluster-randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pharmacist Intervention Arm (Experimental): Pharmacist to prescribe/monitor/manage oral anticoagulation therapy for atrial fibrillation stroke prophylaxis (under collaborative practice agreement with participants primary care provider) in accordance with ACC/AHA/HRS Guidelines.
  Interventions: Drug: Oral anticoagulant
- Enhanced Usual Care Control Arm (Active Comparator): Pharmacist to notify primary care provider that patient has 'actionable' atrial fibrillation and provide current medication list.
  Interventions: Drug: Oral anticoagulant

INTERVENTIONS:
Drug: Oral anticoagulant — Anticoagulant therapy will be initiated/titrated in patients with atrial fibrillation in accordance with ACC/AHA/HRS Guidelines
  Other Names: warfarin; novel oral anticoagulants

SUMMARY:
This is a prospective, open-label, cluster-randomized controlled trial of 400 participants (aged 60 years or older, with additional stroke risk factors and 'actionable' undertreated AF) from a total of 40 retail and outpatient community pharmacies. Participants will be randomized (by pharmacy) to either to an intervention arm of pharmacist-led OAC management versus an enhanced usual care arm, wherein physicians receive notification of 'actionable' AF and patients are advised to schedule a physician clinic visit. The primary objective will be to determine the difference in proportion of patients with 'actionable AF' receiving guideline concordant OAC therapy at 3 months in those randomized to intervention arm versus control arm.

DETAILED DESCRIPTION:
Oral anticoagulation therapy for stroke prevention in AF is safe and effective but under-utilized. Optimal delivery of existing therapies would prevent AF-related stroke. Therefore alternative strategies to increase adherence to current guidelines for OAC use for AF stroke prevention should be explored.

Accumulating data indicate that pharmacist-led or pharmacist-collaborative care in cardiovascular disease monitoring, risk factor control, and medication optimization leads to greater adherence to guideline-directed targets and improved outcomes.

In this prospective, open-label, cluster-randomized controlled trial the investigators intend to enroll 400 participants (aged 60 years or older, with additional stroke risk factors and 'actionable' undertreated AF) from a total of 40 retail and outpatient community pharmacies in Los Angeles. Participants will be randomized (by pharmacy) to either to an intervention arm of pharmacist-led OAC management versus an enhanced usual care arm, wherein physicians receive notification of 'actionable' AF and patients are advised to schedule a physician clinic visit. The primary objective will be to determine the difference in proportion of patients with 'actionable AF' receiving guideline concordant OAC therapy at 3 months in those randomized to intervention arm versus control arm. Secondary outcomes include: patient satisfaction with pharmacist services (at 3 months), pharmacists' perspective on study implementation (at study end), and OAC adherence (at 1 year). In an exploratory aim, the investigators will assess healthcare utilization and clinical outcomes at 1 year.

This research will generate new knowledge on an innovative, and potentially sustainable stroke prevention strategy to increase evidence-based use of OAC therapy in patients with AF.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 60 years
2. Men (CHADS-VASc score ≥2) AND Women (CHADS-VASc score ≥3)
3. AF and not on OAC therapy but eligible
4. AF and on sub-optimal or inappropriate OAC therapy
5. Written informed consent

Exclusion Criteria:

1. AF on optimal OAC therapy
2. OAC required for other conditions (i.e. DVT/PE, PCI in prior year, left ventricular thrombus, etc.)
3. Currently taking two antiplatelet agents
4. Uncontrolled hypertension (defined as SBP ≥160 mmHg x 2 BP readings measured at screening)
5. End-stage renal disease (CrCl <15 ml/min or dialysis)
6. Major surgery in prior month (defined as surgery requiring general anesthesia and overnight inpatient hospital stay)
7. History of "major bleeding" in prior year (defined as overt bleeding at critical site including intracranial, intraspinal, intraocular, pericardial, GI bleed, bleed requiring hospitalization, bleed resulting in ≥20 g/L drop in hemoglobin or requiring transfusion of ≥2 units packed cells)
8. Excess alcohol intake (≥8 alcoholic drinks/week)
9. Inability to read or understand English or Spanish
10. Participants considered unreliable by the Investigator or designated pharmacy team member concerning the requirements of follow-up, or those with foreshortened life expectancy precluding 3-month follow-up
11. Severe cognitive impairment (≥5 errors on the Short Portable Mental Status Questionnaire)
12. Pregnant women

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Optimal OAC Therapy | At 3 months
  To determine the difference in proportion of patients with 'actionable AF' receiving optimal OAC therapy at 3 months in those randomized to intervention arm versus control arm.

SECONDARY OUTCOMES:
'Actionable' AF Prevalence | Through study completion, an average of 1 year
  To determine the prevalence of patients with 'actionable AF'
Medication Adherence (NOAC) | At 12 months
  To assess OAC adherence (i.e. proportion of days covered (PDC) for NOACS)
Medication Adherence (Warfarin) | At 12 months
  To assess OAC adherence (i.e. time in the therapeutic range (TTR) for warfarin)
Patient Satisfaction with Pharmacist Services | At 3 months
  To assess patient satisfaction with pharmacist services using 22-item questionnaire
Qualitative Review of Program Implementation | Through study completion, an average of 1 year
  To perform a qualitative review of program implementation by surveying pharmacists about their experiences with 11-item questionnaire
Healthcare Utilization | At 12 months
  To assess healthcare utilization (i.e. the number of physician visits, specialist visits, ED visits, and hospitalizations)

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No